CLINICAL TRIAL: NCT03148028
Title: Immunological Characteristics of Patients With Primary Immunodeficiencies and Inflammatory Bowel Diseases
Brief Title: Immunological Characteristics of Patients With PID and IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-17-3824-DS-CTIL
Record Dates: First submitted 2017-04-27; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Inflammatory Bowel Diseases; Primary Immune Deficiency Disorder
MeSH Terms: conditions — Inflammatory Bowel Diseases; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — PBMCs Serum Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PID IBD patients: patients with an immunodeficiency and inflammatory bowel disease phenotype

SUMMARY:
The investigators wish to characterize alterations in the architecture and function of immune cells in patients with a primary immunodeficiency that also develop inflammatory bowel disease. In addition, The investigators' goal is to characterize the microbiome of these patients, in order to determine whether specific microbial alterations are related to inflammation.

DETAILED DESCRIPTION:
The pathogenesis of inflammatory bowel diseases (IBD), like Crohn's disease and ulcerative colitis is complex and is thought to be related to genetic, environmental and microbial alterations that lead to a hyperactive/dysregulated immune system that mediates tissue damage. In rare cases, IBD can develop in patients with primary immunodeficiencies (PID) who develop severe, atypical or recurrent infections. The bowel disease in these patients can present after they develop infectious complications but also prior to that. The goal of the current study is to characterize immune function in patients with PID and IBD in order to identify alterations in pro-inflammatory and regulatory pathways.

The investigators will obtain blood samples from PID patients with IBD in order to perform deep immune profiling using various techniques such as flow cytometry, ELISA and others. Moreover, the investigators wish to characterize the microbiome of these patients. This multi-disciplinary approach will advance our understanding why specific patients with an immunodeficiency develop an IBD-like phenotype.

ELIGIBILITY:
Inclusion Criteria:

* age <18 years
* diagnosis of an immunodeficiency
* suspected or confirmed IBD

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a known or unknown immunodeficiency who develop inflammatory bowel disease or are suspected to have such a condition.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of immune cells | 3 years
  Frequency of pro- and anti-inflammatory immune cell subsets including functional analysis

SECONDARY OUTCOMES:
Characterization of stool microbiome | 3 years
  16S analysis to identify changes in diversity and specific taxa

CONTACTS AND LOCATIONS:
Overall Officials: Dror S Shouval, MD, Principal Investigator — Edmond and Lily Safra Children's Hospital
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Be'er Sheba
  - Edmond and Lily Safra Children's Hospital, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No